CLINICAL TRIAL: NCT05371834
Title: Pivotal Study to Assess the Clinical Efficacy and Safety of Microwave Treatment in Warts
Brief Title: Microwave Treatment of Common and Plantar Warts
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Blackwell Device Consulting (Industry)
Collaborators: Emblation Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EMBHPV02
Record Dates: First submitted 2022-05-05; First posted 2022-05-12 (Actual); Last update posted 2024-05-21 (Actual); Status verified 2024-05

CONDITIONS: Warts
Keywords: HPV; Human Papilloma Virus; Swift System; Microwave; Verruca; Common warts; Plantar Warts; Cryotherapy
MeSH Terms: conditions — Warts | interventions — Cryotherapy

STUDY DESIGN:
Masking Description: This is an open label study, however, there is a blinded site investigator at each site who will not be aware of the treatment group the subject is assigned. The blinded site investigator will assess resolution and reoccurrence of the warts. Photos of the warts will be taken and these will be reviewed by three independent blinded assessors to assess wart resolution and reoccurrence.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Microwave Treatment (Swift System) (Experimental): 5-10 Watts of microwave energy applied locally on each wart for a 2-3 second burst with 3-5 repetitions per lesion.
  Interventions: Device: Microwave Treatment (Swift System)
- Cryotherapy Treatment (Active Comparator): For each wart, two cycles of cryotherapy treatment is administered.
  Interventions: Device: Cryotherapy

INTERVENTIONS:
Device: Microwave Treatment (Swift System) — Localized microwave energy applied to the wart lesion. Treatment is in 4-week intervals (minimum of 2 treatments, maximum of 4 treatments).
  For common warts (usually hands, elbow, knees): Treatment starts at 6W and applied locally for a 2 second burst and the dose and duration is adjusted (up or down) as is tolerable for the subject. Treatment is repeated on the same wart as is tolerable (3-5 repetitions).
  For plantar warts: Treatment starts at 8W and applied locally for a 2 second burst and the dose and duration is adjusted (up or down) as is tolerable for the subject. Treatment is repeat on the same wart as is tolerable (3-5 repetitions).
  Less power for a longer time will result in a more gradual temperature rise. Higher power for a shorter time will result in a more immediate temperature rise.
  Arms: Microwave Treatment (Swift System)
Device: Cryotherapy — Local application of Cryotherapy. Treatment is in 4-week intervals (minimum of 2 treatments, maximum of 4 treatments).
  Arms: Cryotherapy Treatment

SUMMARY:
This is a multi-center, open, randomized, parallel-group, controlled, blind-assessed trial of approximately 124 subjects that require treatment for up to 5 common or plantar warts. Subjects will be randomized to one of two treatment groups: Microwave Treatment (Swift® system) or Cryotherapy.

DETAILED DESCRIPTION:
The primary objective of this study is to collect evidence of the effectiveness of the Swift device for the treatment of common and plantar warts and compare with Cryotherapy.

The secondary objectives of this study are to collect evidence of the safety, effectiveness and patient experiences of the Swift device for the treatment of common and plantar warts and compare with Cryotherapy.

Eligible subjects who provide written informed consent will be randomized to either Microwave Treatment or Cryotherapy. Each eligible subject will receive treatment at the baseline visit (Visit 2) and again 4-weeks later. Subjects will receive a minimum of 2 treatments or, if further treatment is required, up to a maximum of 4 treatments; each treatment is given in 4-week intervals. Follow-up is 12-weeks after the last treatment has been administered where the warts will be assessed for resolution. Further follow-up visits occur 6-months and 12-months after the last treatment where the warts will be assessed for resolution or reoccurrence (if resolved at the 12-week visit).

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated informed consent form;
2. Stated willingness to comply with all study procedures and availability for the duration of the study;
3. Age 18-64 years inclusive;
4. A minimum of one clinically significant common wart (usually found on hands, knees and elbows), or one plantar wart. Note: the warts for treatment cannot be a mixture of common and plantar warts;
5. Subject's common warts must measure between 3mm-10mm or for plantar warts, measure between 3mm-20mm, inclusive;
6. If currently receiving treatment for common or plantar warts, agree to stop their current medication for at least 28 days prior to the start of study treatment;
7. Agrees to refrain from using any other wart removal products or treatments during the study period;
8. Agrees to not take any non-steroidal anti-inflammatory drugs (NSAIDs) or antihistamines within a 12-hour period prior to and after randomized treatment;
9. Able to perform study assessments.

Exclusion Criteria:

1. Pregnancy or breast feeding;
2. Mosaic warts for treatment;
3. Warts (common or plantar) that have been reported by the subject as present for more than 5 years (relates to any wart present and which may not necessarily be treated in this study);
4. Warts for treatment on areas of thin or sensitive skin as determined by the Investigator, e.g., face, neck, armpits, breasts, buttocks or genitals;
5. Areas for treatment where the skin is irritated, reddened or showing any sign of inflammation (e.g. itching and swelling);
6. Warts for treatment with hair growth, birthmarks, dark moles, pigmented skin or any other unusual skin condition;
7. History of infection in designated treatment area within 90 days prior to first treatment;
8. Implantable Cardioverter Defibrillator (ICD), pacemaker or other implantable electronic devices;
9. Metal implants at site of treatment (within foot or ankle);
10. Known allergy or intolerance to microwave therapy and cryotherapy;
11. Unstable co-morbidities (cardiovascular disease, active malignancy, inflammatory arthritis);
12. Participating in another interventional study or have done so within the last 30-days;
13. Anticipated relocation or extensive travel outside of the local study area preventing compliance with study procedures;
14. Circulatory conditions affecting the acral areas - peripheral vascular disease, peripheral ischemia, vasculitis, Raynaud's, or related conditions;
15. Peripheral neuropathy;
16. Subject with known immunosuppression disorders through illness or medication (for example - corticosteroids, biologic agents, methotrexate, ciclosporin);
17. Subject with autoimmune disease;
18. Diabetes (Type I or II);
19. History of vascular interventions to the legs, deemed as an unacceptable risk by the Investigator;
20. Prior dissection of axillary lymph nodes (for treated hand) or inguinal lymph nodes (for treated feet);
21. Dependent lymphedema;
22. Congestive heart failure;
23. History of repeated cellulitis (2 or more episodes);
24. History of deep venous thrombosis;
25. Subject currently receiving prescribed blood thinning medication;
26. Subject who has ever had any topical metallic treatment (e.g, aluminum chloride, silver nitrate) within the past year.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 119 (Actual)
Dates: Start 2022-07-06 (Actual); Primary Completion 2024-08 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
Clearance of all treated warts, each of which is defined as "resolved" or "not resolved" based on the classification by the blinded site investigator assessing the treated warts at three months post final treatment (up to 5 warts in total). | 3 months post final treatment

SECONDARY OUTCOMES:
Clearance of all treated warts at three months post final treatment, each of which is defined as "lesion no longer visible" but assessed by the majority of three independent blinded assessors using photographs | 3 months post final treatment
Efficacy of all warts classed as resolved by the blinded site investigator at three months post final treatment, by the number of warts treated | 3 months post final treatment
Patient reported satisfaction with treatment at six and twelve months post final treatment | 6 and 12 months post final treatment
  A patient reported satisfaction questionnaire will be completed. The questionnaire relates to how satisfied the subject was about their treatment and likes/ dislikes about their treatment.
Adverse events | 12 months post final treatment
Change from baseline for size of treated warts at three months, six months and at twelve months post final treatment | 3 months, 6 months and 12 months post final treatment
Patient reported pain score since last treatment at three, six and twelve months post final treatment | 3 months, 6 months and 12 months post final treatment
  The subject will be asked to rate the worst pain they have experienced (None, Mild, Moderate, Severe).
Reoccurrence of any treated wart at six and twelve months post final treatment, as classified by the blinded site investigator and separately by photos reviewed by the majority of the three independent blinded assessors. | 6 months and 12 months post final treatment
Clearance of all treated warts, each of which is defined as "resolved" or "not resolved" based on the classification by the blinded site investigator assessing the treated warts at six months and twelve months post final treatment. | 6 months and 12 months post final treatment
The resolution rate for individual warts based on the classification by the blinded site investigator at 3 months post-final treatment. | 3 months post final treatment

CONTACTS AND LOCATIONS:
Overall Officials: Dr Bhatia, Principal Investigator — Oak Dermatology
Locations (6):
- United States (6):
  - Miami Dermatology and Laser Institute, Miami, Florida
  - TrueBlue Clinical Research, Palm Harbor, Florida
  - TrueBlue Clinical Research, Tampa, Florida
  - Weil Foot & Ankle Institute, Chicago, Illinois
  - Oak Dermatology, Naperville, Illinois
  - Tennessee Clinical Research Center, Nashville, Tennessee